CLINICAL TRIAL: NCT02051504
Title: Impact of Type 1 Diabetes and Glycated Haemoglobin Levels on Oxygen Delivery and Release to Active Muscle During Exercise and on Muscle Oxidation Capacity - Possible Impact on Aerobic Fitness
Brief Title: Muscle Oxygenation, Type 1 Diabetes, and Glycated Hemoglobin
Acronym: OXYDIAB
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2009_12; 2009-A00746-51. (Other: ID-RCB number, AFSSAPS)
Record Dates: First submitted 2013-12-20; First posted 2014-01-31 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; Glycated hemoglobin; Muscle Oxygenation; Exercise; Maximal Oxygen uptake; Mitochondrial respiration; Endocannabinoid system; Oxidative stress
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity | interventions — Glucose Tolerance Test; Absorptiometry, Photon; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, plasma, serum, and skeletal muscle (vastus lateralis) samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Type 1 diabetes, HbA1c <7%: Patients with Type 1 diabetes and adequate glycemic control: HbA1c <7% at the entrance in the study.
  Intervention:
  Incremental maximal exercise Near-Infra Red-Spectroscopy at vastus lateralis and pre-frontal cortex (during exercise) Gas exchanges (VO2, VCO2) during exercise Combined DLCO/DLNO (at rest) Venous and arterialised blood sampling (rest and exercise) Muscle biopsy at the vastus lateralis (rest) Diet questionnaire, quality-of-life questionnaires, physical activity questionnaires Accelerometry over one week Dual energy X-ray Absorptiometry
  Interventions: Behavioral: Incremental maximal exercise; Procedure: Muscle biopsy; Procedure: Combined DLCO-DLNO; Procedure: Dual energy X-ray absorptiometry; Procedure: Accelerometry over one week; Other: Questionnaires
- Type 1 diabetes, HbA1c >8%: Patients with Type 1 diabetes and inadequate glycemic control: HbA1c >8% at the entrance in the study.
  Intervention:
  Incremental maximal exercise Near-Infra Red-Spectroscopy at vastus lateralis and pre-frontal cortex (during exercise) Gas exchanges (VO2, VCO2) during exercise Combined DLCO/DLNO (at rest) Venous and arterialised blood sampling (rest and exercise) Muscle biopsy at the vastus lateralis (rest) Diet questionnaire, quality-of-life questionnaires, physical activity questionnaires Accelerometry over one week Dual energy X-ray Absorptiometry
  Interventions: Behavioral: Incremental maximal exercise; Procedure: Muscle biopsy; Procedure: Combined DLCO-DLNO; Procedure: Dual energy X-ray absorptiometry; Procedure: Accelerometry over one week; Other: Questionnaires
- Healthy controls, Groupe 1: Healthy controls for patients with Type 1 diabetes and adequate glycemic control matched on age, sex, body composition and physical activity level.
  Intervention:
  Oral Glucose Tolerance Test Incremental maximal exercise Near-Infra Red-Spectroscopy at vastus lateralis and pre-frontal cortex (during exercise) Gas exchanges (VO2, VCO2) during exercise Combined DLCO/DLNO (at rest) Venous and arterialised blood sampling (rest and exercise) Muscle biopsy at the vastus lateralis (rest) Diet questionnaire, quality-of-life questionnaires, physical activity questionnaires Accelerometry over one week Dual energy X-ray Absorptiometry
  Interventions: Behavioral: Incremental maximal exercise; Dietary Supplement: Oral Glucose Tolerance Test; Procedure: Muscle biopsy; Procedure: Combined DLCO-DLNO; Procedure: Dual energy X-ray absorptiometry; Procedure: Accelerometry over one week; Other: Questionnaires
- Healthy controls, Group 2: Healthy controls for patients with Type 1 diabetes and inadequate glycemic control matched on age, sex, body composition and physical activity level.
  Intervention:
  Oral Glucose Tolerance Test Incremental maximal exercise Near-Infra Red-Spectroscopy at vastus lateralis and pre-frontal cortex (during exercise) Gas exchanges (VO2, VCO2) during exercise Combined DLCO/DLNO (at rest) Venous and arterialised blood sampling (rest and exercise) Muscle biopsy at the vastus lateralis (rest) Diet questionnaire, quality-of-life questionnaires, physical activity questionnaires Accelerometry over one week Dual energy X-ray Absorptiometry
  Interventions: Behavioral: Incremental maximal exercise; Dietary Supplement: Oral Glucose Tolerance Test; Procedure: Muscle biopsy; Procedure: Combined DLCO-DLNO; Procedure: Dual energy X-ray absorptiometry; Procedure: Accelerometry over one week; Other: Questionnaires

INTERVENTIONS:
Behavioral: Incremental maximal exercise — The exercise test starts 2-4h after a standardised breakfast. After a 2-min resting period sitting on the cycle ergometer (Excalibur Sport, Lode B.V, Medical Technology, Groningen, Netherlands), the test starts at 30 watts with a 20 watts increment every 2min until exhaustion.
Dietary Supplement: Oral Glucose Tolerance Test — The subjects arrive after an overnight fast and have a 75g Glucose Oral Charge.
  Groups: Healthy controls, Group 2; Healthy controls, Groupe 1
Procedure: Muscle biopsy — A sample of vastus lateralis (less than 150mg) is taken with a specific needle under local anesthesia.
Procedure: Combined DLCO-DLNO — Lung carbon monoxide and nitric oxide diffusion capacities are assessed at rest in a sitting position.
Procedure: Dual energy X-ray absorptiometry — Body composition is measured using dual energy X-ray absorptiometry at rest.
Procedure: Accelerometry over one week — The subjects wear an uniaxial accelerometer over one week to assess their usual physical activity level
Other: Questionnaires — Diet questionnaire, quality-of-life questionnaires, physical activity questionnaires

SUMMARY:
Most of the studies concerning aerobic fitness in Type 1 diabetic patients noted a relationship between impaired aerobic fitness and high glycated haemoglobin (HbA1c) levels, reflecting poor long term glycaemic control. To explain this relationship, the indirect effect of chronically high blood glucose levels on cardiovascular complications - and hence on exercise cardiovascular adaptations - are often mentioned. However, one could wonder if HbA1c could also have a direct impact on aerobic fitness patients with Type 1 diabetes. Haemoglobin glycation may increase its O2 affinity, thus limiting the O2 availability at the muscular level and impairing maximal aerobic power. Moreover, chronic hyperglycaemia might have deleterious effect on muscle mitochondrial capacity to use O2. The aim of this study is to assess the effect of Type 1 diabetes and of HbA1c level on muscular oxygen delivery and use and hence on aerobic fitness.

DETAILED DESCRIPTION:
The current study aims at assessing the impact of Type 1 diabetes and HbA1c on muscle oxygen delivery and on muscle mitochondrial capacity. Our hypothesis is that these both steps of the oxygen cascade might be involved in the aerobic fitness impairment usually observed in poor-controlled patients.

Adults with Type 1 diabetes, aged 18-40 years, without microvascular and macrovascular diabetic complications, will be recruited among patients that regularly attend the unit of diabetology of the University Hospital of Lille and the regional hospital of Roubaix. They will be separated into 2 groups according to their glycaemic control at entrance in the study (HbA1c < 7%, HbA1c > 8%). Subsequently, two healthy control groups (checked by an OGTT) will be selected to strictly match the patients with Type 1 diabetes (age, sex, BMI, number of hours of physical activity per week, tobacco smoking). This is a cross-sectional study including 4 groups.

On their first visit, after the determination of HbA1c, all the subjects will perform at rest a DLCO/DLNO. Then they will realise an incremental exercise test to exhaustion on an electromagnetic cycle ergometer. Non-invasive measures will be performed throughout the exercise test, including gas exchange parameters (and maximal oxygen uptake), muscular and brain oxygenation (Near Infra Red Spectroscopy at vastus lateralis muscle and at prefrontal cortex). A blood sample from an arterialised ear-lobe will be taken at rest and exhaustion to determine O2 haemoglobin saturation, arterial partial pressure in O2 and CO2, haemoglobin concentration, hematocrit, and bicarbonates. Blood, from a catheter in a superficial cubital vein, will also be taken at rest, at a precise time during the exercise and immediately after the exercise to measure potential of hydrogen, bicarbonates, haemoglobin concentration, hematocrit, erythrocyte 2,3-diphosphoglycerate, and other blood markers of metabolic and hormonal adaptations to exercise. The subjects will also fill in questionnaires.

On a second visit, in a fasting state, the subjects will have a muscle biopsy at vastus lateralis using a specific needle (less than 150mg) in order to assess mitochondrial respiration capacity and endocannabinoid system activity. A venous blood sampling will allow analysing other health markers (lipid profile, insulin resistance...).

On another visit, the subjects will have a measure of body composition by Dual energy X-ray Absorptiometry and skinfold thickness.

They will also wear an accelerometer over one week and fill in a diet questionnaire over 3 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 1 diabetes (duration of Type 1 diabetes > 1 year and < 20 years)
* Healthy subjects

Exclusion Criteria:

Exclusion Criteria for patients with Type 1 diabetes:

* Maturity onset diabetes of the young, mitochondrial diabetes, Type 2 diabetes
* Macro or microvascular complications of diabetes

Exclusion Criteria for healthy controls :

• Diabetes (Glycaemia > 11 mmol/L two hours after the OGTT)

Exclusion Criteria for all subjects :

* Obesity (Body Mass Index > 30 kg/m2)
* Contra-indication to maximal exercise
* Pregnant or breast-feeding women
* Other chronic disease than diabetes
* Muscle or articular problems

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The two groups of patients with Type 1 diabetes are recruited from primary care clinics (university hospital of Lille and hospital of Roubaix, France) among patients with Type 1 diabetes for more than 1 year and free from micro and macrovascular complications.
  Healthy participants are selected from a list (n=250) drawn up from patients' friends and contacts. Each healthy control is chosen to strictly match a patient with type 1 diabetes according to gender, age, physical activity levels, and tobacco status.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2010-03; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Maximal oxygen uptake | Participants will perform the incremental maximal exercise on visit 1, one week minimum and 8 weeks maximum after their inclusion in the protocol
  Incremental maximal exercise with gas exchange measure

SECONDARY OUTCOMES:
Arterial oxygen content during maximal exercise | Prior to the incremental maximal exercise on visit 1, and immediately after the incremental maximal exercise on visit 1.
  measured in ear-lobe arterialised capillary samples
Oxyhemoglobin dissociation at active muscle during maximal exercise | On visit 1, continuously during the incremental maximal exercise
  Deoxyhemoglobin and total hemoglobin assessed at vastus lateralis by Near Infrared Spectroscopy
Mitochondrial respiration capacity of vastus lateralis muscle | Participants will have a muscle biopsy on visit 2, performed 3 days minimum and 32 weeks maximum after their visit 1.
  Vastus lateralis muscle sample is obtained by the percutaneous technique after local anesthesia. The mitochondrial respiration is then studied in situ in saponin-skinned fibers.
Prefrontal cortex oxygenation during exercise | On visit 1, continuously during the incremental maximal exercise
  Total hemoglobin and oxyhemoglobin are assessed at the left prefrontal cortex using Near-Infrared Spectroscopy.

OTHER OUTCOMES:
Other factors than hemoglobin glycation that could influence arterial oxygen content | Prior to the incremental maximal exercise on visit 1
  Lung capillary carbon monoxide and nitric oxide diffusion capacities (DLCO, DLNO)
Other factors able to modify the oxyhemoglobin dissociation curve | Prior to the incremental maximal exercise on visit 1, and immediately after the incremental maximal exercise on visit 1.
  venous erythrocyte 2,3-diphosphoglycerate, arterialised capillary potential of hydrogen oxygen partial pressure, carbon dioxide partial pressure
Mechanisms possibly involved in muscle mitochondrial dysfunctions | Prior to the incremental maximal exercise on visit 1, and immediately after the incremental maximal exercise on visit 1. Prior to the muscle biopsy on visit 2.
  oxidative stress (blood oxidative and antioxidant markers at rest and in response to maximal exercise), endocannabinoid system activity
Other health markers in link with physical activity levels and aerobic fitness | Prior to the incremental maximal exercise on visit 1, and immediately after the incremental maximal exercise on visit 1. Prior to the muscle biopsy on visit 2.
  Lipid profile (HDL-C, LDL-C, apolipoprotein A1, apolipoprotein B, lipoprotein a, ...) Insulin resistance markers (blood ghrelin, adiponectin, leptin...)
Blood metabolic and hormonal responses to exercise | Prior to the incremental maximal exercise on visit 1, and immediately after the incremental maximal exercise on visit 1.
  Free fatty acids, glycerol, glucose, insulin, catecholamines, glucagon, cortisol, insulin-like growth factor 1, brain-derived neurotrophic factor...
Body composition | Prior to incremental maximal exercise on visit 1
  Dual energy X-ray Absorptiometry, skinfold thickness, waist and hip circumferences

CONTACTS AND LOCATIONS:
Overall Officials: Elsa HEYMAN, PHD, Study Director — EA4488 'Physical activity, Muscle, Health; Pierre FONTAINE, MD-PHD, Principal Investigator — CHRU LILLE
Locations (1):
- CHRU Lille, Lille, France

REFERENCES:
- [Derived] Jlali I, Heyman E, Matran R, Marais G, Descatoire A, Rabasa-Lhoret R, Touil I, Pawlak-Chaouch M, Mucci P, Fontaine P, Baquet G, Tagougui S. Respiratory function in uncomplicated type 1 diabetes: Blunted during exercise even though normal at rest! Diabet Med. 2023 May;40(5):e15036. doi: 10.1111/dme.15036. Epub 2023 Jan 10. PMID 36585956
- [Derived] Lespagnol E, Tagougui S, Fernandez BO, Zerimech F, Matran R, Maboudou P, Berthoin S, Descat A, Kim I, Pawlak-Chaouch M, Boissiere J, Boulanger E, Feelisch M, Fontaine P, Heyman E. Circulating biomarkers of nitric oxide bioactivity and impaired muscle vasoreactivity to exercise in adults with uncomplicated type 1 diabetes. Diabetologia. 2021 Feb;64(2):325-338. doi: 10.1007/s00125-020-05329-8. Epub 2020 Nov 21. PMID 33219433
- [Derived] Heyman E, Daussin F, Wieczorek V, Caiazzo R, Matran R, Berthon P, Aucouturier J, Berthoin S, Descatoire A, Leclair E, Marais G, Combes A, Fontaine P, Tagougui S. Muscle Oxygen Supply and Use in Type 1 Diabetes, From Ambient Air to the Mitochondrial Respiratory Chain: Is There a Limiting Step? Diabetes Care. 2020 Jan;43(1):209-218. doi: 10.2337/dc19-1125. Epub 2019 Oct 21. PMID 31636081
- [Derived] Tagougui S, Fontaine P, Leclair E, Aucouturier J, Matran R, Oussaidene K, Descatoire A, Prieur F, Mucci P, Vambergue A, Baquet G, Heyman E. Regional cerebral hemodynamic response to incremental exercise is blunted in poorly controlled patients with uncomplicated type 1 diabetes. Diabetes Care. 2015 May;38(5):858-67. doi: 10.2337/dc14-1792. Epub 2015 Feb 9. PMID 25665816
- [Derived] Tagougui S, Leclair E, Fontaine P, Matran R, Marais G, Aucouturier J, Descatoire A, Vambergue A, Oussaidene K, Baquet G, Heyman E. Muscle oxygen supply impairment during exercise in poorly controlled type 1 diabetes. Med Sci Sports Exerc. 2015 Feb;47(2):231-9. doi: 10.1249/MSS.0000000000000424. PMID 24983346